CLINICAL TRIAL: NCT00490945
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Study of the Effects of VEC-162 on Circadian Rhythm in Healthy Subjects
Brief Title: Safety and Efficacy of VEC-162 on Circadian Rhythm in Healthy Adult Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VP-VEC-162-2101
Record Dates: First submitted 2007-06-22; First posted 2007-06-25 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: Circadian Rhythm Sleep Disorders
MeSH Terms: conditions — Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: VEC-162

SUMMARY:
The purpose of this study is to assess the safety and efficacy of VEC-162 compared to matching placebo on circadian phase shift and sleep parameters.

ELIGIBILITY:
Inclusion Criteria:

* No medical, psychiatric, or sleep disorders
* Ability to provide written informed consent

Exclusion Criteria:

* Lifetime history of night shift work
* Evidence of any sleep disorder
* Psychiatric or neurological disorders

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2004-07; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marlene Dressman, PhD, Study Director — Vanda Pharmaceuticals Inc
Locations (2):
- United States (2):
  - Vanda Investigational Site, Boston, Massachusetts
  - Vanda Investigational Site, Detroit, Michigan

REFERENCES:
- [Derived] Rajaratnam SM, Polymeropoulos MH, Fisher DM, Roth T, Scott C, Birznieks G, Klerman EB. Melatonin agonist tasimelteon (VEC-162) for transient insomnia after sleep-time shift: two randomised controlled multicentre trials. Lancet. 2009 Feb 7;373(9662):482-91. doi: 10.1016/S0140-6736(08)61812-7. Epub 2008 Dec 4. PMID 19054552

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Number of Enrolled Subjects = 45 Number of Enrollment Failures = 6
Groups:
- Placebo: Randomized to Placebo
- 10 mg VEC-162: Randomized to 10 mg VEC-162
- 20 mg VEC-162: Randomized to 20 mg VEC-162
- 50 mg VEC-162: Randomized to 50 mg VEC-162
- 100 mg VEC-162: Randomized to 100 mg VEC-162
Period: Overall Study
Arm/Group | Placebo | 10 mg VEC-162 | 20 mg VEC-162 | 50 mg VEC-162 | 100 mg VEC-162
Started | 8 | 9 | 8 | 7 | 7
Completed | 8 | 8 | 8 | 7 | 7
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 10 mg VEC-162 | 20 mg VEC-162 | 50 mg VEC-162 | 100 mg VEC-162 | Total
Number analyzed (Participants) | 8 | 9 | 8 | 7 | 7 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.5 (6.7) | 31.8 (7.4) | 32.5 (9.6) | 27.4 (6.2) | 30.4 (9.5) | 30.0 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 4 | 4 | 4 | 20
  Male | 3 | 6 | 4 | 3 | 3 | 19

OUTCOME MEASURES:

1. Primary Outcome: Circadian Phase Shift
Description: Exposure response to VEC-162 on induction of circadian phase shift as measured by Dim Light Melatonin Onset (DLMO) was defined as the time change between Night 3 and Night 4 when melatonin production reached 25% of the maximum melatonin concentration. Samples below LOQ of the melatonin assay were assigned 5 pg/ml.
Time Frame: Night 3 and Night 4
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Placebo | 10 mg VEC-162 | 20 mg VEC-162 | 50 mg VEC-162 | 100 mg VEC-162
Number analyzed (Participants) | 6 | 8 | 7 | 4 | 5
Hours | -0.48 (0.84) | 0.18 (2.48) | -1.14 (0.46) | -0.50 (0.32) | -2.74 (1.95)

2. Primary Outcome: Mean Sleep Efficiency
Description: Exposure response was measured by comparing the change in sleep efficiencies of VEC-162 and placebo treated subjects upon a sleep schedule phase advance. Sleep efficiency (total time asleep divided by the time allowed as an opportunity for sleep in a period multiplied by 100%, where time allowed for sleep was 8 hours or 480 minutes) was measured objectively by overnight polysomnographic recordings. Sleep efficiency was also compared in parts of the night by dividing the full night into thirds.
Time Frame: Night 4 and Night 2
Population: *N = 6 for 3rd Third of Night Efficiency and N=8 for 1st Third of Night Efficiency
  **N = 7 for 3rd Third of Night Efficiency
Measure: Mean (Standard Deviation); unit: % points
Groups:
- Placebo*: Randomized to Placebo
- 10 mg VEC-162: Randomized to 10 mg VEC-162**
Arm/Group | Placebo* | 10 mg VEC-162 | 20 mg VEC-162 | 50 mg VEC-162 | 100 mg VEC-162
Number analyzed (Participants) | 7 | 8 | 8 | 7 | 7
% points
  Full Night (% points) | -20.27 (18.72) | -7.77 (14.98) | -6.68 (12.69) | -5.87 (9.89) | -2.02 (4.94)
  1st Third of the Night (% points) | -12.30 (14.51) | -0.47 (12.39) | -7.81 (14.52) | 0.95 (7.79) | -5.63 (17.71)
  2nd Third of the Night (% points) | -34.92 (38.23) | -12.64 (13.83) | -5.11 (12.78) | -2.10 (4.14) | -2.30 (5.72)
  3rd Third of the NIght (% points) | -8.06 (29.69) | -10.51 (35.17) | -7.09 (26.24) | -16.48 (26.25) | 1.80 (14.15)

3. Secondary Outcome: Wake After Sleep Onset (WASO), and Latency to Persistent Sleep (LPS)
Description: Wake After Sleep Onset is defined as the total time that is scored as awake in a PSG occurring between sleep onset and lights-on prompt.
  Latency to Persistent Sleep is defined as the number of epochs (one 30-second interval of the sleep episode) from the beginning of the recording (lights-out) to the start of persistent sleep (first 20 consecutive non-wake state) divided by 2.
Time Frame: Night 2 and Night 4
Population: *Placebo N = 7 and 100 mg VEC-162 N = 7
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | 10 mg VEC-162 | 20 mg VEC-162 | 50 mg VEC-162 | 100 mg VEC-162
Number analyzed (Participants) | 8 | 8 | 8 | 7 | 6
minutes
  Latency to Persistent Sleep | 15.13 (21.25) | -8.25 (16.34) | 5.00 (11.89) | -3.71 (10.97) | -4.17 (6.93)
  WASO* | 77.00 (91.01) | 40.56 (67.53) | 31.19 (53.80) | 31.21 (52.69) | 8.50 (20.39)

4. Secondary Outcome: VEC-162 AUC
Time Frame: Night 4
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | 10 mg VEC-162 | 20 mg VEC-162 | 50 mg VEC-162 | 100 mg VEC-162
Number analyzed (Participants) | 9 | 8 | 7 | 7
ng*hr/mL | 171.73 (118.51) | 482.00 (329.48) | 614.34 (488.08) | 1916.06 (601.35)

5. Secondary Outcome: VEC-162 Cmax
Time Frame: Night 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 10 mg VEC-162 | 20 mg VEC-162 | 50 mg VEC-162 | 100 mg VEC-162
Number analyzed (Participants) | 9 | 8 | 7 | 7
ng/mL | 59.10 (39.22) | 139.94 (116.10) | 166.01 (164.94) | 417.80 (187.19)

6. Secondary Outcome: VEC-162 Tmax
Time Frame: Night 4
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | 10 mg VEC-162 | 20 mg VEC-162 | 50 mg VEC-162 | 100 mg VEC-162
Number analyzed (Participants) | 9 | 8 | 7 | 7
hour | 1.90 (1.78) | 2.04 (0.90) | 2.42 (0.59) | 3.03 (1.50)

ADVERSE EVENTS:
Time Frame: 1st dose to 30 days following last administration of study treatment
Arm/Group | Placebo | 10 mg VEC-162 | 20 mg VEC-162 | 50 mg VEC-162 | 100 mg VEC-162
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/8 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 8/8 | 8/9 | 7/8 | 7/7 | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=8) | 10 mg VEC-162 (N=9) | 20 mg VEC-162 (N=8) | 50 mg VEC-162 (N=7) | 100 mg VEC-162 (N=7)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival Hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal Tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Application Site Irritation (General disorders) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Injection Site Pain (General disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Injection Site Bruising (General disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Application Site Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Feeling Hot (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Application Site Reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection Site Anaesthesia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection Site Burning (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection Site Discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection Site Erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection Site Irritation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection Site Movement Impairment (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes Simplex (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematocrit Decreased (Investigations) | 3 (3) | 4 (4) | 3 (3) | 4 (4) | 4 (4)
Haemoglobin Decreased (Investigations) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 3 (3)
Blood Pressure Systolic Decreased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Blood Pressure Diastolic Decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood Pressure Diastolic Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutrophil Count Decreased (Investigations) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood Phosphorus Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Potassium Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Pressure Systolic Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Electrocardiogram Abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eosinophil Count Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart Rate Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Heart Rate Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Lymphocyte Count Increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Monocyte Count Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Platelet Count Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 4 (7) | 3 (3) | 2 (3) | 5 (7) | 2 (2)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (3)
Dizziness (Nervous system disorders) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 1 (2)
Syncope Vasovagal (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Nervousness (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abnormal Dreams (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mental Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep Disorder (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal Discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No